CLINICAL TRIAL: NCT02362607
Title: Integrated Diabetes Management Protocol Using Smartphone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chungbuk National University (Other)
Responsible Party: Principal Investigator, Hyung Jin Choi, Clinical Assistant Professor, Chungbuk National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-06-006
Record Dates: First submitted 2015-02-02; First posted 2015-02-13 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

ARMS (2):
- Integrated Diabetes Management Protocol (Experimental): Smartphone apps for food diary, activity monitor, blood glucose will be used for three months.
  Interventions: Behavioral: Integrated Diabetes Management Protocol
- Standard Diabetes Management Protocol (Active Comparator): Subjects will receive standard diabetes management protocol with standard education and standard blood glucose measurement devices.
  Interventions: Behavioral: Standard Diabetes Management Protocol

INTERVENTIONS:
Behavioral: Integrated Diabetes Management Protocol
  Arms: Integrated Diabetes Management Protocol
Behavioral: Standard Diabetes Management Protocol
  Arms: Standard Diabetes Management Protocol

SUMMARY:
The investigators aim to assess whether using integrated diabetes management protocol using smartphone would increase glucose control among diabetes patients.

DETAILED DESCRIPTION:
Smartphones and digital healthcare is expected to provide better diabetes care. The investigators aim to assess whether using integrated diabetes management protocol using smartphone would increase glucose control among diabetes patients.

Smartphone apps for food diary, activity monitor, blood glucose will be used for three months.

Blood glucose control and patient satisfaction will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, type 1 diabetes, gestational diabetes

Exclusion Criteria:

* Medications which interfere glucose control
* Cancer
* Chronic kidney injury

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Blood Glucose Control Status Measured by HbA1c | After three months
  Blood test results for HbA1c after three months.

SECONDARY OUTCOMES:
Patient Satisfaction Measured by Questionnaire | After three months
  Summary of Diabetes Self-Care Activities Measure (SDSCA) Questionnaire (Toobert et al., 2000)

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University, Cheongju-si, North Chungcheong, South Korea